CLINICAL TRIAL: NCT04156984
Title: Exposure-response of Golimumab During Maintenance in Ulcerative Colitis: An Exploratory Pharmacokinetics/Pharmacodynamics Comparison of Different Dose Regimens
Brief Title: Comparison of Two Different Golimumab Dosing Regimens for Ulcerative Colitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: David Drobne (Other)
Responsible Party: Sponsor-Investigator, David Drobne, Principal investigator, University Medical Centre Ljubljana
Organization: University Medical Centre Ljubljana (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-001G
Record Dates: First submitted 2019-10-24; First posted 2019-11-08 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Ulcerative Colitis
Keywords: Pharmacokinetics; Pharmacodynamics; Safety; Golimumab; Reactive dose optimisation; Proactive dose optimisation; Golimumab concentration; Mucosal healing; Therapeutic drug monitoring; Inflammatory bowel disease; Personalized medicine; Comparisons of European with US label
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Study arm (Other): Subjects treated with optimized dose of golimumab, irrespective of weight: golimumab 200 mg sc, followed by 100 mg sc at week 2 and then 100 mg sc q4 weeks. In case of disease flare: discontinuation of drug.
  Interventions: Drug: Golimumab Prefilled Syringe
- Control arm (Other): Subjects treated according to current European Label (2019) based on body weight:
  1. <80kg: golimumab 200 mg sc, followed by 100 mg sc at week 2 and then 50 mg sc q4wk. In case of disease flare (defined as PRO-2 ≥1): dose optimization to 100 mg sc q4wk starting at week 6 or at any time during first year.
  2. ≥80kg: golimumab 200 mg sc, followed by 100 mg sc at week 2 and then 100 mg sc q4wk. In case of disease flare (defined as PRO-2 ≥1): discontinuation of drug.
  Interventions: Drug: Golimumab Prefilled Syringe

INTERVENTIONS:
Drug: Golimumab Prefilled Syringe — See arm description

SUMMARY:
Partial response or loss of response to golimumab is observed in a significant proportion of patients started on golimumab for active ulcerative colitis. The current dosing regimen in European Union is based on patients' body weight as maintenance treatment for patients with ≥ 80 kg is 100 mg q4 weeks and for patients with <80 kg 50 mg q4 weeks. The investigators recent observations in a golimumab pharmacokinetics study of 24 patients however, show large interindividual variations in golimumab trough concentrations. Furthermore, it seems that patients with continuous response have higher golimumab trough levels at several time points during treatment compared to patients who lose response. Higher induction/maintenance dose of golimumab increases golimumab trough levels, therefore it is likely that higher induction/maintenance dose of golimumab would increase efficacy of golimumab treatment.

DETAILED DESCRIPTION:
Partial response or loss of response to golimumab is observed in a significant proportion of patients started on golimumab for active ulcerative colitis. The current dosing regimen in European Union is based on patients' body weight as maintenance treatment for patients with ≥ 80 kg is 100 mg q4 weeks and for patients with <80 kg 50 mg q4 weeks. The investigators recent observations in a golimumab pharmacokinetics study of 24 patients however, show large interindividual variations in golimumab trough concentrations. Furthermore, it seems that patients with continuous response have higher golimumab trough levels at several time points during treatment compared to patients who lose response. Higher induction/maintenance dose of golimumab increases golimumab trough levels, therefore it is likely that higher induction/maintenance dose of golimumab would increase efficacy of golimumab treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed ulcerative colitis

Exclusion Criteria:

* Active tuberculosis or other opportunistic bacterial, viral and fungal infections
* History of moderate to severe heart failure (NYHA III/IV), and potential risk of congestive heart failure
* Pregnancy
* History of allergic reactions to sorbitol (E420), L-histidine, L-histidine monohydrochloride monohydrate, polysorbate80, water for injections.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2021-04-07 (Actual); Primary Completion 2024-06-18 (Actual); Study Completion 2024-06-18 (Actual)

PRIMARY OUTCOMES:
Endoscopic outcome | 50 weeks
  Number of participants with mucosal healing at week 14 and week 50 on flexible rectosigmoidoscopy (recorded and assessed centrally by blinded reader if possible). Mucosal healing is defined as Mayo endoscopic score 0 or 1.

SECONDARY OUTCOMES:
Clinical outcome | 50 weeks
  Number of participants in clinical remission at week 14, week 26, week 38 and week 50. Clinical remission is defined as PRO-2 (Patient-Reported Outcome) score 0 (no rectal bleeding and no diarrhea/altered bowel habit).
Association of golimumab through levels and Anti-golimumab antibodies development on endoscopic and clinical outcome. | 50 weeks
  Measurement of golimumab through levels. Blood withdrawals will be preformed at prespecified time points in all patients: week 0, week 2, week 4, week 6, week 10, week 14, week 26, week 38 and week 50.
  Measurement of Anti-golimumab antibodies development. Blood withdrawals will be preformed at prespecified time points in all patients: week 2, week 4, week 6, week 10, week 14, week 26, week 38 and week 50.

OTHER OUTCOMES:
Measurement of physical, social, and emotional status with The Short Inflammatory Bowel Disease Questionnaire. | 50 weeks
  The Short Inflammatory Bowel Disease Questionnaire (SIBDQ) is a health-related quality of life (HRQoL) tool measuring physical, social, and emotional status (score 10-70, poor to good HRQoL). The questionnaire will be answered at week 0, week 6, week 14, week 26, week 38, week 50.
Incidence of Treatment-Emergent Adverse Events as assessed by CTCAE v4.0. | 50 weeks.
  Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0.

CONTACTS AND LOCATIONS:
Overall Officials: David Drobne, MD, PhD, Principal Investigator — University Medical Centre Ljubljana; Borut Štabuc, MD, PhD, Study Director — University Medical Centre Ljubljana
Locations (4):
- Slovenia (4):
  - General hospital Celje, Department of Gastoenterology, Celje
  - General hospital Izola, Department of Internal medicine, Izola
  - University Medical Centre Ljubljana, Department of Gastroenterology, Ljubljana
  - University Medical Centre Maribor, Department of Gastoenterology, Maribor

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Stefanovic S, Detrez I, Compernolle G, Brouwers E, Sever N, Stabuc B, Smrekar N, Kurent T, Novak G, Kozelj M, Ferrante M, Gils A, Drobne D. Endoscopic remission can be predicted by golimumab concentrations in patients with ulcerative colitis treated with the changed label. Eur J Gastroenterol Hepatol. 2021 Jan;33(1):54-61. doi: 10.1097/MEG.0000000000001843. PMID 32804854